CLINICAL TRIAL: NCT06966050
Title: Multi-center MRD Registry for Inflammatory Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-0415; NCI-2025-03109 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2025-04-25; First posted 2025-05-11 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Participants will fill out a quality-of-life questionnaire and complete a MRD test.
  Interventions: Behavioral: Quality-of-life Questionnaire

INTERVENTIONS:
Behavioral: Quality-of-life Questionnaire — Participants will be asked to fill out a quality-of-life questionnaire, which will take about 10-15 minutes to complete.

SUMMARY:
To collect data from participants with IBC who may have had MRD testing and may have surgery in the future.

DETAILED DESCRIPTION:
Primary Objectives

-To determine the incidence of protocol specified pre-surgery MRD-positivity in IBC (assessment between completion of planned systemic therapy and surgery).

Secondary Objectives

* To establish the feasibility of multi-institutional MRD data collection using standard of care Signatera analysis in IBC participants.
* To evaluate the association of pre-surgery MRD to pathologic response.
* To evaluate participant reported QOL for worry about recurrence based in participants receiving MRD results
* To establish protocol-optional baseline and longitudinal MRD data collection in IBC participants and report the frequency of MRD longitudinally
* To determine the median lead time between the first MRD-positive result and clinical recurrence.
* To determine whether adjuvant therapies decrease the amount of MRD in participants, and the association with relapse.

ELIGIBILITY:
Inclusion Criteria:

* Female or males ≥18 years of age with the ability to understand and sign a written
* Participants who have a clinical diagnosis of stage III or IV inflammatory breast cancer (IBC).
* Participants who are planning to have or already completed a minimum of one blood draw for Signatera testing, for which the result and clinical data can be deposited into the study database.
* Participants must be within eight months of diagnosis and have not undergone breast surgery for this diagnosis of breast cancer.
* Participants must be English-speaking.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2030-05-31 (Estimated); Study Completion 2032-05-31 (Estimated)

PRIMARY OUTCOMES:
European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire | Through study completion; an average of 1 year
  European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30)
  Score scale: (1-30 questions to assess the impact of participants quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Sadia Saleem, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2025-04-24): https://cdn.clinicaltrials.gov/large-docs/50/NCT06966050/ICF_000.pdf